CLINICAL TRIAL: NCT01837732
Title: Effectiveness of Relational Touch in the Management of Chronic Pain in Institutionalized Elderly
Brief Title: Effectiveness of Relational Touch in Painful Elderly
Acronym: EFFITOUREL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K110702; 2012-AO1042-41 (Other: IDRCB)
Record Dates: First submitted 2013-04-02; First posted 2013-04-23 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Pain
Keywords: Chronic pain; elderly; relational touch
MeSH Terms: conditions — Chronic Pain | interventions — Relational Autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: relational touch (Experimental): Relational touch 15 mn " relational touch", hand touch (neck, face and head)
  Interventions: Other: Relational Touch
- B: relational (Active Comparator): Relational: 10 mn verbal patient's centered exchanges
  Interventions: Other: Relational:

INTERVENTIONS:
Other: Relational Touch — Relational touch 15 mn " relational touch", hand touch (neck, face and head)
  Arms: A: relational touch
Other: Relational: — Relational: 10 mn verbal patient's centered exchanges
  Arms: B: relational

SUMMARY:
The aim is to investigate the feasibility and efficacy of a relational touch / relational intervention on persistent pain in a long term geriatric hospital care ward population. The main issue is the pain reduction. The hypothesis is that this type of intervention is very useful on pain reduction in old people even with physical or mental disability.

DETAILED DESCRIPTION:
The first 74 patients wanting to participate are randomly assigned to 2 groups: relational- touch or relational. Inclusion criteria are : patients with chronic pain; age >65y and informed consent. Where patients had mental impairment the family's agreement is solicited. The regional Ethics Committee agreement was granted. The intervention consists of 6 Relational versus Relational- Touch sessions (twice a week) .Evaluation takes place after the second, 4th and 6th sessions and in the 4th week following the intervention. The main outcome is the pain reduction.

The primary outcome measure is the pain reduction according to the DOLOPLUS scale and the VRS; the secondary outcomes measures are : patient's participation rate; pain related symptoms variation; overall benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 y
* Chronic pain > 3 months
* Follow up 4 weeks
* Patient's speak french
* Patient's or representative's agreement to participate and to the informatics treatment of the data

Exclusion Criteria:

* acute pain
* unstable clinical status

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
SCALE DOLOPLUS BEHAVIORAL ASSESSMENT OF PAIN IN THE ELDERLY (DOLOPLUS pain score variations) | change from baseline to 4th week
  Pain assessment : DOLOPLUS pain score variations at baseline and in the 4th week following the intervention (for all patients)

SECONDARY OUTCOMES:
Scale of Guy (Pain related symptoms) | at 3th week and 4th week
  Pain related symptoms variation at 3th week (session 6) and 4th week (session 9)(for all patients)
Global benefit questionary | 2 sessions per week for 4 weeks and one after the 6 sessions
  Global benefit : 2 sessions per week for 4 weeks and one after the 6 sessions following the intervention (for all patients)
Acceptability rate at each session | 2 sessions per week for 3 weeks and in 4 th week
  Acceptability rate at each session and proportion of the patients completing the whole treatment (for all patients)
score variations of Verbal Rating Scale (VRS) | change from baseline to 4th week
  Pain variation according to VRS at baseline and in the 4th week following the intervention (for communicative patients only)
Global benefit questionary (nurse, doctor, carer) | after the 6 sessions
  Global benefit : 2 after the 6 sessions following the intervention by nurse, doctor, carer for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Philippe JOSEPH-SYLVESTRE, Nurse, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital René Muret - Head of department Long Term hospital ward, Sevran, France